CLINICAL TRIAL: NCT01278667
Title: Difficulties in Emotional Processing, the Influence of Methylphenidate on This Processing and the Relations Between Emotional Processing and Social Functioning Among Children With ADHD
Brief Title: Methylphenidate and the Relations Between Emotional Processing and Social Functioning Among Children With ADHD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Bnai Zion Medical Center (Other Government)
Responsible Party: Roni Geva, Dept of Psychology, Fac of Social Sciences, Bar Ilan University, Ramat Gan, Israel
Other Study IDs: 80-10-BNZ
Record Dates: First submitted 2011-01-16; First posted 2011-01-19 (Estimated); Last update posted 2011-01-25 (Estimated); Status verified 2011-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; Memory; Social; Emotion; Methylphenidate
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Children with ADHD are in high risk to develope social difficulties. The present study will examine the emotional processing in those children. The main purpose is to investigate the connection between memory and recognition of facial expressions, how those abilities influence social functioning and if Methylphenidate influence the emotional processing.

The study will include 80 children in ages 9-12 years, devided in 2 groups; children with ADHD treated with Methylphenidate, and healthy children without ADHD. The children will do computerized tasks that examine recognition and memory of facial expressions. Social function will be examined by questionnaires filled by parents and teachers.

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity Disorder (ADHD) is characterized by short attention and concentration, impulsive and hyperactive behavior. Children with ADHD are in high risk to develop difficulties in social adjustment. The social difficulties challenge the support that those children get from their environment through their lives.

Last years studies on the causes that influence ADHD's social difficulties, suggests that they derive from problems in emotional information processing. Some research focus on recognition deficits of emotion and facial expressions, but their results are inconsistent. Moreover, there is a disagreement about the problems in the emotional processing that influence the social behavior of children with ADHD.

In the present study we will further examine the emotional information processing in children with ADHD. We will focus on recognition and memory of facial expressions. The main purpose of the current study is to investigate the connection between memory and recognition of facial expressions, and how those abilities influence social functioning. Another purpose is to investigate the assumption that beyond impulsivity and inattention, the difficulty in emotional processing is caused by specific deficits in the capacity to recognize and recall facial expressions. In order to test this assumption we will compare between the ability to recognize and recall facial expressions and the ability to recognize and recall objects.

ADHD is positively influenced by arousing drugs. Methylphenidate is the most prescribed and investigated drug in Israel. This drug improves attention, social and cognitive functions, and reduces hyperactive and impulsive behavior. However, its influence on emotional processing was not studied enough. Another purpose of this study is to test the efficiency of this drug on emotional processing.

The present study will include 80 children in ages 9-12 years, divided in 2 groups; 40 children with ADHD treated with Methylphenidate, and 40 healthy children without ADHD. The ADHD group will be tested in 2 sessions; one under drug treatment and one without drug treatment. The healthy children will be tested in 1 session. The children will do computerized tasks (Complex Reaction Time, Modified Day-Night and Attention Network Test) that examine recognition and memory of facial expressions. In order to examine their social function, their parents and teachers will fill questionnaires (BRIEF, CBCL/6-18 and TRF/6-18).

ELIGIBILITY:
Inclusion Criteria:

* children with ADHD under treatment with methylphenidate

Exclusion Criteria:

* non-cooperative children
* children suffering from other neurological or mental conditions
* children suffering from asthma

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children with ADHD are in high risk to develope social difficulties. The present study will examine the emotional processing in those children. The main purpose is to investigate the connection between memory and recognition of facial expressions, how those abilities influence social functioning and if Methylphenidate influence the emotional processing.
  The study will include 80 children in ages 9-12 years, recruited from a community sample include schools in Haifa. They will devided in 2 groups; children with ADHD treated with Methylphenidate, and healthy children without ADHD. The children will do computerized tasks that examine recognition and memory of facial expressions. Social function will be examined by questionnaires filled by parents and teachers.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2011-01; Primary Completion 2011-12 (Estimated); Study Completion 2012-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Schwartz, MD, Principal Investigator — Dep. of Neurology, Bnai Zion Medical Center, Haifa, Israel
Locations (1):
- Dep. of Neurology, Bnai Zion Medical Center, Haifa, Israel